CLINICAL TRIAL: NCT03651193
Title: Multi-center Registration Study of Adult Onset Still's Disease in Chinese Population
Acronym: MAOSDC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Qianjin Lu, MD, PhD, Professor and Director, Dept. of Dermatology, The Second Xiangya Hospital of Central South University, Second Xiangya Hospital of Central South University
Other Study IDs: MAOSDC20180720
Record Dates: First submitted 2018-08-27; First posted 2018-08-29 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Adult Onset Still Disease
Keywords: Adult Onset Still's Disease; Chinese population
MeSH Terms: conditions — Still's Disease, Adult-Onset

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — whole blood 5ml，serum 1.5ml
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AOSD: Patients fulfill Japan's Yamaguch AOSD classification
  Interventions: Diagnostic Test: Exon sequencing and Methylated sequencing
- Control: Use 1:1 group matching, should meet the following condition -s : same gender as matching case; same age as matching case or the difference ranges within 1 year; no Immune related diseases (e.g. Psor -iasis, Systemic Lupus Erythematos -us, Dermatomyositis, Scleroderma, Rheumatoid Arthritis, Type 1 Diabet -es, Behcet's disease, Sjogren's Syndrome, Hyperthyroidism, etc.); no family history of immune related diseases.
  Interventions: Diagnostic Test: Exon sequencing and Methylated sequencing

INTERVENTIONS:
Diagnostic Test: Exon sequencing and Methylated sequencing — Exon sequencing and Methylated sequencing

SUMMARY:
This multi-center registration study will investigate the clinical characteristics of AOSD population in China , identify possible factors inducing the onset and active condition of AOSD in Chinese population , and identify the new high specific and sensitive markers of AOSD

DETAILED DESCRIPTION:
Backgrounds: Adult-onset Still's disease (AOSD) is a rare systemic clinical syndrome of unknown etiology. Its pathogenesis is complex, often thought to be affected by infection, genetic and immune factors. Due to the low incidence of adult Still's disease and the lack of specific clinical features and laboratory tests, infections, tumors, connective tissue diseases and other diseases must be excluded before clinical diagnosis. Therefore, the diagnosis of adult Still's disease is still a great challenge for clinicians at this stage. Moreover, the process of exclusion diagnosis is long, and examinations, including some invasive examinations, are bringing heavy burden to the patients psychologically, physiologically and economically.

The clinical manifestations of AOSD vary greatly, and AOSD is typically characterised by spiking fever, arthritis, evanescent rash. Other non-specific symptoms may be observed in AOSD: involvement of lymphatic/reticuloendothelial system can cause sore throat, lymph node enlargement; involvement of respiratory and cardiovascular system can cause chest pain and dyspnea; involvement of the liver can cause liver enlargement and abnormal liver function. In addition, it can involve all major systems of the body. Common laboratory indicators include: WBC> 10 000 / mm3, with neutrophils> 80%, abnormal increased erythrocyte sedimentation rate (ESR) and C-reactive protein (90% - 100% in AOSD), Hyperferritinemia ( specificity of 80%) and IL-18 (sensitivity of 91.7% and specificity of 99.1%). However, both clinical symptoms and laboratory examinations are not unique to the disease, and infections, tumors, connective tissue diseases and so on often exhibit similar characteristics. Therefore, these diseases need to be excluded before the diagnosis of adult Still's disease in order to prevent delays in diagnosis and missing the best opportunity for treatment .

At present, the treatment of AOSD is usually empirical and diagnostic, mainly using NSAIDs, steroids, DMARDS and biological agents. Although these treatments can effectively relieve symptoms and improve the quality of life of patients, but still cannot cure the disease. A small number of patients can be remitted within a year and no longer relapse; about one-third of patients relapse several times in uncertain interval , with lighter symptoms and shorter duration than the initial onset after complete remission ; the rest of the patients will be chronic. Besides, a small number of serious patients will develop into macrophages. Activation syndrome often threatens life. Therefore, most patients need long-term monitoring and even lifelong medication.

At present, there is no national study on AOSD with large sample size in China, and many foreign studies on the potential biomarkers of AOSD still need to be further explored in terms of sensitivity and specificity. The investigators carried out this study to collect at least 150 pairs of clinical data and blood samples from patients with AOSD and age-and sex-matched normal controls through collaboration of multiple units throughout the country, and to perform genome-wide exon sequencing and methylation sequencing in order to identify the genetic and epigenetic characteristics of specific changes in AOSD. On this basis, further studies on pathogenesis are carried out.The results of this study may reveal the main pathogenesis of adult Still's disease, identify potential biomarkers with high sensitivity and specificity in peripheral blood, thus simplifying the diagnostic process, shortening the diagnostic cycle, reducing invasive examinations, alleviating the psychological, physiological and economic burden of patients in the diagnostic process, and providing AOSD with a new direction for diagnosis and treatment.

Design of Study: This is a cross sectional survey and 1:1 case-control study to explore the clinical characteristics of AOSD population in China; Identify possible factors inducing the onset and active condition of AOSD in Chinese population ;Identify new markers of AOSD with high specificity and sensitivity.

Methods: Pre-experiment preparation: design data collection form, determine the final data collection form and experimental plan, establish multiple experimental centers across the country.

After sample screening, informed consent, determine join in this study or not. Divide those population agree to join into AOSD group and Controlled group(1:1 matching). Then carry out Case study, case-control study and disease impact investigation among AOSD group, carry out case-control study and disease impact investigation among controlled group. Case study include investigating characteristics and relationship between AOSD and exposure factors among AOSD group. Case-control study is comprised of study of living environment and dietary exposure, social, and psychological factors ,behavior, genetics, epigenetics, immunology, biomarkers. Disease impact investigation covers Psychological emotion , social burden and quality of life. The results are to analyzed using multivariate logistic regression analysis: overall factors.

ELIGIBILITY:
Inclusion Criteria:

* AOSD: Patients fulfill Japan's Yamaguch AOSD classification.
* Control: Use 1:1 group matching, should meet the following condition -s : same gender as matching case; same age as matching case or the difference ranges within 1 year; no Immune related diseases (e.g. Psor -iasis, Systemic Lupus Erythematos -us, Dermatomyositis, Scleroderma, Rheumatoid Arthritis, Type 1 Diabet -es, Behcet's disease, Sjogren's Syndrome, Hyperthyroidism, etc.); no family history of immune related diseases.

Exclusion Criteria:

* Anyone with physical or mental illness that may affect the assessment will be excluded, such as patients with hearing or speech expression disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Chinese population
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2018-11-28 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
gene expression level and methylation level | 0 day
  The data of this study is managed by the Hunan Key Laboratory of Medical Epigenomics (Department of Dermatology, The Second Xiangya Hospital of Central South University). The authenticity, integrity and confidentiality of clinical data are required to be ensured, original case and case report form shall be filled out by investigator or the designated person of researcher and shall not be altered at will. If necessary, the name of the changer and the date of modification should be signed.
  Statistical analysis will use GraphPad Prism or SPSS software. All statistical tests will be performed using a two-sided test, P values less than 0.05 will be considered statistically significant, the confidence interval uses 95%. The measurement data will be statistically described using mean ± standard deviation or median (minimum, maximum). Disease exposure factors and impact analysis will be based on descriptive statistical analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Qianjin Lu, MD，PHD, Principal Investigator — Central South University
Locations (1):
- The Second Xiangya Hospital of Central South University, Hunan, Changsha, China

IPD SHARING:
Plan to Share IPD: No